CLINICAL TRIAL: NCT00989924
Title: Research on the Correlation Among Magnetocardiography Patterns and Known Cardiovascular Risk Factors in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Lee-Ming Chuang/professor, National Taiwan University Hospital
Other Study IDs: 200906039R
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Coronary heart disease; Magnetocardiography
MeSH Terms: conditions — Diabetes Mellitus; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetes mellitus: The Diabetic patient who receives follow-up at NTUH diabetics caring network

SUMMARY:
The purpose of this study is to evaluate the correlation among magnetocardiography (MCG) patterns and various known cardiovascular risk factors.

DETAILED DESCRIPTION:
It is well understood that diabetes mellitus (DM) causes various micro- and macrovascular complications. Among them, coronary heart diseases (CHDs) claim most mortality, and diabetes has been considered as "CHD equivalent". Furthermore, the risk of CHD has been noticed to increase in the pre-diabetic stage, suggesting the development of CHD may start in a rather early stage of the disease. Thus, early detection of CHD in diabetic patients seems to be important. However, currently exam methods for CHD in diabetic patients seemed to have their limitations.

Developed in the 1960s, magnetocardiography (MCG) is designed to detect the weak magnetic field generated by the electrical activity of the heart, and has been used widely in the study of fetal cardiac electrophysiology, arrhythmia and ischemic heart disease. However, the MCG pattern in diabetic patients is not fully understood. The aim of the study is to clarify the correlation among various cardiovascular risk factors and MCG pattern in diabetic patients. And, according to the results of the study, we'll evaluate the potentiality of MCG in early diagnosis of CHD in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Clear consciousness
* Met the diagnostic criteria of DM published by the American Diabetes Association in 2009

Exclusion Criteria:

* not suitable for MCG exam (ex. with pacemaker implantation or indwelling metallic device)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Diabetic patient who receives follow-up at NTUH diabetics caring network
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2009-10

PRIMARY OUTCOMES:
The smooth index of corrected QT interval (SIQTC) measured by MCG | as the MCG exam is over

CONTACTS AND LOCATIONS:
Overall Officials: Lee-Ming Chuang, MD. Ph.D., Study Director — National Taiwan University Hospital; Chau-Chung Wu, MD. Ph.D., Principal Investigator — National Taiwan University Hospital; Yi-Der Jiang, MD., Principal Investigator — National Taiwan University Hospital; Tien-Jyun Chang, MD. Ph.D., Principal Investigator — National Taiwan University Hospital; Chih-Hung Lin, MD., Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan